CLINICAL TRIAL: NCT01070017
Title: Community-based Accompaniment With Supervised Antiretrovirals in Lima, Peru
Acronym: CASA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Partners in Health (Other); Harvard School of Public Health (HSPH) (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Sonya Sunhi Shin, Dr., Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01MH083550-01A2 (NIH); 1R01MH083550-01A2 (NIH)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: HIV; AIDS; HIV Infections
Keywords: Peru; DOT; HIV; AIDS; Community based; social capital
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Intervention Model Description: Cluster randomization of sites assign individuals starting antiretroviral therapy to receive community-based directly observed therapy plus home visits / social support versus home visits / social support alone.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention: DOT-HAART (Experimental): Intervention group will receive community-based monthly adherence visits, standard care, and DOT-HAART.
  Interventions: Other: DOT-HAART
- No DOT-HAART (No Intervention): Control group receives community-based monthly adherence visits and standard care, but no DOT-HAART.

INTERVENTIONS:
Other: DOT-HAART — For 8 months, DOT-HAART of all doses in the participant's home or alternate location. DOT worker ensures that HIV medications are taken as indicated and witnesses ingestion of all medications including other medications prescribed by physician. The worker will be trained to identify, triage and notify providers of any psychosocial and medical problems/complications. Transition to self-administration begins in months 9-12 when DOT will be tapered and greater participation of treatment supporter to prepare patients for self-administration.
  Arms: Intervention: DOT-HAART

SUMMARY:
Using quantitative and qualitative data, this study will assess the impact of community accompaniment with supervised antiretrovirals (CASA) on HIV-positive individuals and community members in Lima, Peru.

DETAILED DESCRIPTION:
Community-based accompaniment with directly observed antiretroviral therapy (DOT-HAART) may improve adherence and clinical outcomes among impoverished individuals starting HAART in resource-poor settings. Furthermore, the utilization of community health workers may build social capital. This is cluster-randomized trial, with randomization at the level of health centers. Individuals in both intervention and control clusters will receive community-based adherence support (monthly adherence visits) and standard care. In addition, individuals residing in intervention clusters will receive 12 months of community-based DOT-HAART. We will enroll patients as well as community members (health providers, treatment supporters, and community health workers) to assess individual and community-level outcomes.

ELIGIBILITY:
Inclusion Criteria for Patient Cohort:

* Age greater than or equal to 18;
* Diagnosis if HIV and meeting criteria for HAART;
* Lives in poverty;
* EITHER: 1) HAART naïve or 2) starting salvage therapy due to virologic failure;
* Documentation of baseline CD4 cell count and HIV load;
* Residence and receipt of HIV healthcare within the study catchment area

Exclusion Criteria for Patient Cohort:

- Imprisoned or cannot give informed consent.

Inclusion Criteria for Community Cohort:

* Working in a health establishments in study region;
* If health personnel, contracted employee caring for people living with HIV/AIDS.

Exclusion Criteria for Community Cohort:

- Cannot give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1244 (Actual)
Dates: Start 2010-02; Primary Completion 2012-07-31 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Proportion with suppressed HIV viral load after starting HAART among those receiving community-based DOT-HAART versus the control group. | 18 and 24 months

SECONDARY OUTCOMES:
Identify mediating mechanisms of CASA effect on individual outcomes. | 24 months
Identify subgroups who respond best to CASA intervention. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Shin, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Socios En Salud, Lima, Peru